CLINICAL TRIAL: NCT06486571
Title: Development of Innovative Strategies for the Control of Robotic Hand Prostheses Based on High-density Electromyography and Restitution of Sensory Feedback Via Trans-cutaneous Electrical Stimulation
Brief Title: Strategies to Control Robotic Hand Prosthesis Via HD-sEMG and to Restore Sensory Feedback Via TENS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Nazionale Assicurazione contro gli Infortuni sul Lavoro (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CP-PAS-01-23; 528-2023 (Other: Ethics Committee)
Record Dates: First submitted 2024-06-24; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Upper Limb Amputees
Keywords: Upper limb amputation; HD-sEMG; Pattern recognition; Sensory feedback; TENS
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All participants (Experimental)
  Interventions: Other: Electromyography recording with HD-sEMG; Other: Transcutaneous Electrical Nerve Stimulation (TENS)

INTERVENTIONS:
Other: Electromyography recording with HD-sEMG — Measurement of muscle electrical signal with HD-sEMG sensors, training of a pattern recognition classifier for hand gesture recognition, verification and comparison with state of the art.
Other: Transcutaneous Electrical Nerve Stimulation (TENS) — Application of TENS by means of non-invasive superifical electrodes on the stump skin of the participants to restore multimodal somatotopical sensations of mechanoception, nociception and thermoception.

SUMMARY:
Upper limb amputation still causes severe disability today; prostheses currently on the market are able to restore partially to the amputee the lost functionality. In addition to the motor capacity of the limb, prosthetic systems should also aim to restore to the sensory information from the surrounding environment during contact with objects. Therefore, it is important to develop bidirectional prostheses. It is thus apparent that the development of new techniques for decoding the efferent channel, such as high-density surface electromyography, and for encoding of the afferent channel afferent, to return multimodal somatosensory sensations of mechanoception, nociception, and thermoception using TENS, isimportant to improve the patient's use of the prosthesis.

ELIGIBILITY:
Inclusion Criteria:

* Upper limb amputation;
* Stable clinical condition;
* Skin integrity of the stump;
* Age between 18 and 65 years;
* High level of motivation to participate in the study and acceptance of the purpose of the study;
* Signed informed consent document.

Exclusion Criteria:

* Clinical instability;
* Dehiscence of the amputation wound;
* Failure to complete the informed consent;
* State of pregnancy;
* Implanted devices that can interfere with TENS stimulation (e.g. pacemakers);

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-23 (Actual); Primary Completion 2025-12-22 (Estimated); Study Completion 2026-04-22 (Estimated)

PRIMARY OUTCOMES:
Improve gestures decoding by means of HD-sEMG decoding algorithms | through study completion, an average of 2 year through study completion, an average of 2 year
  The performance of HD-sEMG classifiers with variable number of classes will be evaluated in the offline phase in terms of accuracy of classification and F1-Score.
Elicit somatic sensations in amputees | through study completion, an average of 2 year through study completion, an average of 2 year
  The performance of the stimulation strategy will be evaluated in terms of stimulus discrimination accuracy, a parameter that identifies the number of times the subject correctly reports the type of sensation elicited by the experimenter compared to the total number of stimulations performed.

SECONDARY OUTCOMES:
Increase the number of hand grasps to be classfiied | through study completion, an average of 2 year through study completion, an average of 2 year
  To explore the possibility of increasing the number of gestures that can be classified by the developed classification system, compared to the number of gestures that can be reproduced by prosthetic control solutions traditional and to evaluate the intuitiveness in using classifiers to control a polyarticulated prosthesis.
Development of encoding strategies | through study completion, an average of 2 year through study completion, an average of 2 year
  Develop new algorithms for decoding motor intention from the myoelectric signal and new encoding algorithms for the sensory restitution by non-invasive stimulation and to evaluate the intuitiveness of the developed strategies.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Protesi Inail, Budrio, BO, Italy

IPD SHARING:
Plan to Share IPD: No